CLINICAL TRIAL: NCT04948151
Title: A Phase 2b, Multi-Center, Multiple-Dose, Double-Blind, Placebo-Controlled Study to Evaluate the Efficacy and Safety of Sildenafil Cream, 3.6% in Premenopausal Patients With Female Sexual Arousal Disorder (FSAD)
Brief Title: Multi-Center Study to Evaluate the Efficacy and Safety of Sildenafil Cream (3.6%) in Premenopausal Patients With Female Sexual Arousal Disorder
Acronym: RESPOND
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Strategic Science & Technologies, LLC (Industry)
Collaborators: Daré Bioscience, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SST-6006-013
Record Dates: First submitted 2021-06-24; First posted 2021-07-01 (Actual); Last update posted 2021-07-01 (Actual); Status verified 2021-06

CONDITIONS: Female Sexual Arousal Disorder
Keywords: Sexual Disorder; Arousal Disorder; FSAD
MeSH Terms: conditions — Sexual Dysfunction, Physiological | interventions — Sildenafil Citrate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Sildenafil Cream, 3.6% (Experimental)
  Interventions: Drug: Sildenafil
- Placebo Cream (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Sildenafil — Patients will apply 2-gram applications up to 9 times per month.
  Arms: Sildenafil Cream, 3.6%
Drug: Placebo — Patients will apply 2-gram applications up to 9 times per month
  Arms: Placebo Cream

SUMMARY:
This study is looking to minimize side effects, while maintaining and potentially improving the therapeutic benefit to patients suffering from Female Sexual Arousal Disorder by providing a topical preparation of Sildenafil locally to the vulvar-vaginal tissue.

ELIGIBILITY:
Inclusion Criteria - For Patient Eligibility

1. Patient must be a premenopausal woman, 21 years or older.

   a. Transgender individuals assigned a female gender at birth will be permitted to enroll provided they are not currently undergoing hormone treatment, have not undergone gender reassignment surgery and do not intend to for the duration of the study.
2. Patient is fluent in the English language.
3. Patient is capable of understanding and complying with the protocol and agrees to sign the informed consent document.
4. Patient has been in a stable, monogamous, relationship that was secure and communicative, for at least 6 months prior to Visit 1. The relationship is with one sexual partner, who is sexually functional, both psychologically and physically. The partner will be consistent and available throughout the duration of the study.
5. Based on the clinical interview, in their past, patient had experienced 'normal' sexual function for at least 2 years or longer. Patient has had sexual activity at least two times each month during the last 6 months and agrees to have sexual activity at least two times each month for the duration of the study). Sexual activity can include any activity which may result in sexual stimulation or sexual pleasure e.g., intercourse, caressing, foreplay, masturbation, and oral sex.

   a. Patients who have experienced a recent major life stress (e.g., loss of income, death of a family member) or relationship discord that could interfere with sexual activity (except distress related to FSAD) will be excluded.
6. Women of childbearing potential must agree to continue using an acceptable form of birth control during the study and agree to continue to stay on their dose of birth control throughout the duration of the study. Birth control is not required for confirmed same sex couples, couples with confirmed vasectomy or couples with confirmed tubal ligation.

   1. Acceptable forms of birth control include the following: intrauterine system [IUS], progestin and/or estrogen-containing hormonal oral contraceptives, contraceptive patch, contraceptive implant, contraceptive injection, or the copper-containing intrauterine device (IUD). Patients must be using the progestin and or estrogen-containing hormonal oral contraceptives or contraceptive patch for least 6 months prior to Visit 1 without clinically significant complications in the opinion of the Investigator. Patients must be using the IUS, IUD, contraceptive implant, or contraceptive injection for at least 3 months prior to Visit 1 without clinically significant complications in the opinion of the Investigator.
   2. Vaginal forms of contraception such as contraceptive foams/gels, diaphragms, penile or vaginal condoms, contraceptive vaginal rings, and are not considered acceptable methods of birth control in this study.
   3. While latex and polyisoprene condoms are not an acceptable form of contraception, they may be used for the prevention of sexually transmitted infections.
7. Patient has a body mass index (BMI) from 18 to 35 kg/m2, inclusive.
8. Patient has had a Pap smear performed within three years prior to Visit 1 and can provide documentation indicating normal test results (based on current guidelines as published by the U.S. Preventive Services Task Force).

   a. If the patient cannot provide documentation, a Pap smear will be performed at Visit 1.

   Patients with abnormal findings will be excluded from study participation and be referred for follow-up medical care as appropriate.
9. Patient is medically healthy with no clinically significant medical history, physical examination, gynecological history and examination, laboratory profiles (e.g., hematology, urinalysis), vital signs (e.g., uncontrolled hypertension), or ECGs, as deemed by the Investigator.

   1. Patients who have clinically significant ECG abnormalities at Visit 1 as confirmed by the Investigator will be excluded.
   2. Patients with controlled, treated hypertension (<140/90 mmHg) on up to two medications (excluding alpha blockers and nitrates) with a stable dose for the past 6 months will be considered eligible.
   3. Patients with controlled, treated thyroid disease on a stable medication and dose for the past 6 months will be considered eligible. TSH must be within normal range (confirmed by laboratory test).
10. The participant must agree to not use vaginal hormone therapy (e.g., vaginal estrogen, intravaginal prasterone), vaginal or vulvar lubricants, spermicides, creams or gels, contraceptive foams or vaginal douche products throughout the study period.

    1. Women who self-report abnormal physiological vaginal discharge will be excluded until abnormal physiological discharge resolves.
    2. Patients using systemic (transdermal or oral) therapy must be on a stable dose for at least 6 months prior to Visit 1.
11. Patient must have a total score on the FSDS-DAO >18 through visit 4.

Exclusion Criteria - For Patient Eligibility

1. Patient is nursing or pregnant (based on positive serum pregnancy test), wishes to become pregnant or begin nursing during the study period or was pregnant or nursing within 6 months prior to Visit 1.
2. Patient has more than one sexual partner.
3. Patient is postmenopausal (surgically induced or natural) meeting any of the following criteria:

   1. Bilateral oophorectomy.
   2. 12 months of spontaneous amenorrhea
   3. 6 months of spontaneous amenorrhea with serum FSH levels >40mIU/mL (except for those women on hormone replacement therapy)
4. Patient has any disorder or a history of any disorder that may prevent the successful completion of the study in the opinion of the Investigator.
5. Patient has a significant cardiovascular, hepatic, metabolic, renal, respiratory, gastrointestinal, endocrine, immunologic, dermatologic, hematologic, neurologic, genitourinary, or other unstable medical condition that would contraindicate administration of study medication, interfere with study evaluation, limit study participation, or confound the interpretation of study results in the opinion of the Investigator.
6. Patient has a history of unresolved sexual trauma or abuse that is contributing to any sexual dysfunction problem (desire, arousal, orgasm, etc.) as determined by the clinical interview.
7. Patient with any history of active peptic ulcers or clinically significant bleeding disorders.
8. Patient with a history of clitoral priapism or conditions which may predispose them to clitoral priapism (such as sickle cell anemia, multiple myeloma, or leukemia).
9. Patients with a history of myocardial infarction, stroke, or life-threatening arrhythmia within 6 months prior to Visit 1; patients with resting hypotension (BP <90/50 mmHg); or any history of coronary disease causing angina; or congestive heart failure requiring medical intervention; patients with underlying conditions which can be particularly sensitive to the actions of vasodilators including patients with left ventricular outflow obstruction (e.g., aortic stenosis, idiopathic hypertrophic subaortic stenosis) and patients with impaired autonomic control of blood pressure, or for those for which sexual activity is inadvisable due to their underlying cardiovascular status.
10. Patient with a history of hearing loss (unless born completely deaf).
11. Patient has retinitis pigmentosa, even if the patient feels clinically well at the time of Visit 1. Patients with retinitis pigmentosa will be identified by specifically asking whether they have the condition, if there are visual signs and symptoms of the condition (including questioning patients as to whether they have difficulty seeing at night or in low light, and if they have any visual field deficits that indicate a loss of peripheral or central vision), or if there is a family history.
12. Patient has a history of orthostatic hypotension or orthostatic hypotension which is present at Visit 1, defined as a drop in systolic blood pressure ≥ 20 mm Hg, a drop in diastolic blood pressure ≥ 10 mm Hg, an increase in pulse by 20 beats per minute or experiencing lightheadedness or dizziness at 1 or 3 minutes after the change in position from supine to standing.
13. Patient has a primary complaint of anorgasmia, vaginismus, low desire, or any other primary sexual complaint aside from problems with genital arousal, as determined by the clinical interview.
14. Patient has untreated dyspareunia, vulvovaginal infection or inflammation, inflammatory disorders of the vulva or vagina, vestibulodynia, clitorodynia, or symptomatic vulvovaginal atrophy (defined as women having ≤5% of superficial cells on vaginal smear at baseline,
15. Patient has undergone major pelvic or abdominal surgery that may have caused nerve damage, including, vulvectomy, colostomy, cystostomy, hysterectomy and bladder neck suspension.
16. Patients with comorbid conditions that may cause underlying neurological impairment (i.e., Type 1 or Type 2 diabetes, metabolic syndrome, stroke, myasthenia gravis, multiple sclerosis or spinal cord damage) will be excluded.

    a. Patients who are symptomatic of peripheral neuropathy will be excluded.
17. Patients with pelvic nerve damage secondary to trauma will be excluded.
18. With the exception of anxiety and depression, patient has any current and/or previously reported diagnoses of DSM-IV-TR axis I disorders (e.g., schizophrenia, bipolar disorder) including delirium, dementia and amnestic disorders.

    1. Patients diagnosed with anxiety or depression must be controlled, as determined by the Investigator, and if on a medication (i.e., SSRIs, SNRIs, buspirone, bupropion, and benzodiazepines), on a stable dose for at least the past 6 months.
    2. Patients must have a total score <10 indicating mild depression on the Patient Health Questionnaire-8 (PHQ-8, Appendix G) (a screening and assessment instrument for depression).
    3. Patients must have a total score <6 indicating mild anxiety on the Generalized Anxiety Disorder (GAD-7, Appendix H) (a screening and assessment instrument for anxiety).
    4. Patients who have any history of anti-psychotic therapy within the last year will be excluded.
19. Patients that have a history of gynecological cancer or are under active treatment (or recently completed treatment within the last 6 months) for any cancer which in the Investigator's judgement would interfere with the patient's ability to successfully complete the study will be excluded.

    1. Patients who have been previously treated for dysplasia (precancerous changes) may be included as long as the patient received localized treatment (e.g., cryosurgery or laser).
    2. Patients with a history of radiation to the pelvis will be excluded.
20. Patient has any surgical or medical condition that may interfere with the absorption, distribution, metabolism, or excretion of the test article in the opinion of the Investigator.
21. Patient self-reports a history of substance abuse within two years prior to Visit 1 or exhibits signs of current substance abuse based on Investigator judgement.
22. Patient self-reports a history of alcohol abuse in the two years prior to Visit 1 or exhibits signs of current alcohol abuse based on Investigator judgement.
23. Patient has a history of non-arteritic ischemic optic neuropathy (NAION) or any underlying NAION risk factors.
24. Patient whose sexual function was affected (enhanced or worsened) by any medication within 28 days before Visit 1 and at any time prior to the No Drug Run-in Period of the study.
25. Patient is currently receiving treatment or has received treatment within 1 month (28 days) prior to Visit 1 of any of the following medications: guanylate cyclase stimulators (e.g., Riociguat), clonidine, strong CYP3A4 inhibitors, nitric oxide donors, such as organic nitrates or organic nitrites, and alpha blockers.

    a. Patients who are currently receiving treatment or have received treatment in the past 3 months for FSAD symptoms, pharmacologic (e.g., PDE5 inhibitors in any form except Sildenafil Cream, 3.6% or other experimental therapies used to enhance the arousal response) or non-pharmacologic treatment (e.g., sex therapy), will also be excluded.
26. Patient has positive findings from the urine drug screen (e.g., amphetamines, barbiturates, cocaine, methadone, and opiates). Patients who test positive for amphetamines but are being treated for ADHD with a confirmed legal prescription will be allowed to participate.
27. Patient has positive findings for sexually transmitted infection (gonorrhea, trichomoniasis, chlamydia), and human immunodeficiency virus (HIV) antibodies.
28. Patient reports having an outbreak (blisters, warts, or vesicles) due to any of the following sexually transmitted diseases: genital herpes or HPV at any time point in the past three months.
29. Patient has participated in any clinical research study evaluating another investigational drug or therapy within 30 days before Visit 1 (or 6 half-lives of the investigational agent, whichever is longer) and agrees not to participate in another clinical research study throughout the duration of the study.
30. Patient has any clinically significant abnormal findings on vulvar-vaginal examination performed during the physical and gynecological exams at Visit 1 (e.g., genital skin breaks, irritation, dermatoses, or lesions).
31. Patient currently has moderate to severe current vaginitis, a vaginal infection including bacterial vaginosis, a yeast infection or the presence of yeast based on the Nucleic Acid Amplification (NAAT).

    1. If the patient has a vaginal infection or a positive test for yeast during the screening visit, they may be treated, and the screening visit rescheduled.
    2. If the patient develops a vaginal infection following enrollment into the study, study drug will be withheld, and the patient will be treated for the infection. If the infection cannot be resolved within two weeks the patient will be withdrawn from the study. Treatment of vaginal infections will be allowed twice following enrollment. If the patient develops a third vaginal infection they will be withdrawn from the study.
32. Patient has a pelvic or urinary tract infection.

    1. If the patient has a urinary tract infection during the screening visit, they may be treated, and the screening visit rescheduled.
    2. If the patient develops a urinary tract infection following enrollment into the study, study drug will be withheld, and the patient will be treated for the infection. If the infection cannot be resolved within two weeks the patient will be withdrawn from the study. Treatment of urinary tract infections will be allowed twice following enrollment. If the patient develops a third urinary tract infection they will be withdrawn from the study.
33. Patient self-reports a known hypersensitivity or adverse reaction to any ingredients in the Investigational Product (IP).
34. The patient is an immediate family member, a study site employee, or is in a dependent relationship with a study site employee or anyone who is involved in the conduct of the study (e.g., spouse, parent, child, sibling) or may consent under duress.

Min Age: 21 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 440 (Estimated)
Dates: Start 2021-06-28 (Estimated); Primary Completion 2021-12-15 (Estimated); Study Completion 2021-12-15 (Estimated)

PRIMARY OUTCOMES:
SFQ28 (AS) - 28 Day Recall | SFQ28 score at the end of the Single-Blind Placebo Run-In to the end of the 12-Week Double-blind Dosing period.
  Evaluating the efficacy of Sildenafil Cream, 3.6% measured by change from baseline to end of study in the Arousal-Sensation Domain of the SFQ28.
FSDS-DAO (Q14) - 28 Day Recall | Q14 score at the end of the Single-Blind Placebo Run-In to the end of the 12-Week Double-blind Dosing period.
  Evaluating the efficacy of Sildenafil Cream, 3.6% measured by change from baseline to end of study in the score for feeling concerned by difficulties with sexual arousal - Item #14 only of the FSDS-DAO.

SECONDARY OUTCOMES:
Arousal Diary (SSE) | measured by daily prompt within 24hrs after each sexual event during the Single-Blind Placebo Run-In compared to the last 4 weeks of the Double-Blind Dosing Period.
  Evaluating the efficacy of Sildenafil Cream, 3.6% measured by change from baseline to end of study in the number of Satisfactory Sexual Events, question #11 in teh ARousal Diary.

CONTACTS AND LOCATIONS:
Locations (51):
- United States (51):
  - Coastal Clinical Research, Mobile, Alabama
  - Precision Clinical Trials-Arizona, Phoenix, Arizona
  - Visions Clinical Research -Tucson, Tucson, Arizona
  - Collaborative Neuroscience Network, Garden Grove, California
  - NRC Research Institute, Orange, California
  - Medical Center for Clinical Research - San Diego, San Diego, California
  - Schuster Medical Research Institute, Sherman Oaks, California
  - Downtown Women's Healthcare, Denver, Colorado
  - Coastal Connecticut Research, LLC, New London, Connecticut
  - Intimmedicine Specialists, Washington D.C., District of Columbia
  - South Florida Medical Research, Aventura, Florida
  - AMR Fort Myers, Fort Myers, Florida
  - Clinical Neuroscience Solutions-Orlando, Jacksonville, Florida
  - New Age Medical Research Corporation, Miami, Florida
  - Suncoast Clinical Research - Pasco County, New Port Richey, Florida
  - Healthcare Clinical Data, Inc., North Miami, Florida
  - CNS Healthcare, Orlando, Florida
  - Comprehensive Clinical Research, LLC, West Palm Beach, Florida
  - AGILE Clinical Research Trials, Atlanta, Georgia
  - iResearch Atlanta, Decatur, Georgia
  - Rosemark Women Care Specialists, Idaho Falls, Idaho
  - Great Lakes Clinical Trials, Chicago, Illinois
  - Cypress Medical Research Center, Wichita, Kansas
  - Southern Institute for Women's Sexual Health, Covington, Louisiana
  - Praetorian Pharmaceutical Research, Marrero, Louisiana
  - Boston Clinical Trials, Boston, Massachusetts
  - Women's OB-GYN, P.C. dba Saginaw Valley Medical, Saginaw, Michigan
  - Quality Clinical Research, Omaha, Nebraska
  - Omaha OB GYN Associates, P.C., Omaha, Nebraska
  - Essential Women's Health Associates, Las Vegas, Nevada
  - Office of Doctor Rex G. Mabey Junior, Las Vegas, Nevada
  - Women's Health Research Center, Lawrenceville, New Jersey
  - New Jersey Urology - Bloomfield, Millburn, New Jersey
  - The Center for Specialized Women's Health, Morristown, New Jersey
  - Suffolk Obstetrics and Gynecology, Port Jefferson, New York
  - Velocity Clinical Research - Cleveland (Rapid Medical Research), Cleveland, Ohio
  - Aventiv Research, inc., Columbus, Ohio
  - University Hospitals Landerbrook, Mayfield Heights, Ohio
  - Rivus Wellness & Research Institute, Oklahoma City, Oklahoma
  - Velocity Clinical Research, Providence, Warwick, Rhode Island
  - Coastal Carolina Research Center, North Charleston, South Carolina
  - ClinSearch, Chattanooga, Tennessee
  - Clinical Neuroscience Solutions - Memphis, Memphis, Tennessee
  - Medical Research Center of Memphis, Memphis, Tennessee
  - Urology Associates - Nashville, Nashville, Tennessee
  - TMC Life Research, Houston, Texas
  - Maximos Obstetrics and Gynecology, League City, Texas
  - Clinical Trials of Texas, San Antonio, Texas
  - Health Research of Hampton Roads, Inc., Newport News, Virginia
  - Tidewater Clinical Research, Norfolk, Virginia
  - Seattle Women's Health Research - Gynecology, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Johnson I, Thurman AR, Cornell KA, Symonds T, Hatheway J, Friend DR, Goldstein A. Comparisons and correlations of 1-month recall vs 24-hour recall in patient-reported outcomes of an exploratory, phase 2b, randomized, double-blind, placebo-controlled clinical trial of sildenafil cream, 3.6% for the treatment of female sexual arousal disorder. J Sex Med. 2024 Sep 3;21(9):787-792. doi: 10.1093/jsxmed/qdae086. PMID 39059373
- [Derived] Johnson I, Thurman AR, Cornell KA, Hatheway J, Dart C, Brainard CP, Friend DR, Goldstein A. Preliminary Efficacy of Topical Sildenafil Cream for the Treatment of Female Sexual Arousal Disorder: A Randomized Controlled Trial. Obstet Gynecol. 2024 Aug 1;144(2):144-152. doi: 10.1097/AOG.0000000000005648. Epub 2024 Jun 18. PMID 38889431